CLINICAL TRIAL: NCT07388992
Title: Investigating Specific Gait Patterns in Individuals Living With Multiple Sclerosis
Acronym: GAIT-MS
Status: Not yet recruiting | Type: Observational
Sponsor: SYSNAV (Industry)
Responsible Party: Sponsor
Other Study IDs: PR5030-119; 2025-A02511-48 (Other: ANSM)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis; Healthy Adult
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- people living with Multiple Sclerosis
- Healthy Adult

SUMMARY:
The study aims to investigate specific ambulation patterns characteristic of the quality of gait in people with MS (pwMS)

ELIGIBILITY:
Inclusion Criteria:

For people living with multiple sclerosis (pwMS):

1. Age at inclusion between =18 and =65 years old
2. Signed informed consent and ability to comply with study and follow-up.
3. Confirmed MS diagnosis according to McDonald criteria (2017)
4. Expanded Disability Status Scale EDSS = 6
5. Stable treatment for 2 months before inclusion (for both disease modifying and symptomatic therapies)
6. Ability and willingness to participate in and comply with all study procedures defined in the protocol
7. Subject will be eligible for enrollment in this study only if either affiliated to, or a beneficiary of a social security category

For Healthy volunteers :

1. Age at inclusion between =18 and =65 years old
2. Signed informed consent and ability to comply with study and follow-up.
3. Ability and willingness to participate in and comply with all study procedures defined in the protocol
4. Subject will be eligible for enrollment in this study only if either affiliated to, or a beneficiary of a social security category

Exclusion Criteria:

For pwMS:

1. Participants with a relapse within the past 3 months before the inclusion
2. Participants with significant cognitive disorders, limiting the understanding of the exercises to be performed or presence of apparent communication difficulties hindering the correct collection of data, as assessed by the investigator
3. Past or present pathology other than MS or surgery or trauma impacting gait, ambulatory function or upper limb function, as assessed by the investigator
4. Vulnerable adults: individuals subject to a legal protection measure (guardianship, limited guardianship, or judicial protection) or unable to express their consent.

For healthy volunteers (HV):

1. Participants with significant cognitive disorders, limiting the understanding of the exercises to be performed or presence of apparent communication difficulties hindering the correct collection of data, as assessed by the investigator
2. Past or present pathology or surgery or trauma impacting gait, ambulatory function or upper limb function, as assessed by the investigator
3. Vulnerable adults: individuals subject to a legal protection measure (guardianship, limited guardianship, or judicial protection) or unable to express their consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MS will be recruited from the CHU Lille. Patients will be informed of this study by the Investigator during routine follow-up visits.
  The Investigator will also connect with local patient organizations and share a flyer. This flyer will also be displayed within the Neurology and Neurological Rehabilitation departments of the hospital and diffused to the hospital staff.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ambulation pattern description | enrollment
  ambulation pattern in people living with multiple sclerosis with different disease severities

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Vermersch, Principal Investigator — CHU Lille